CLINICAL TRIAL: NCT02224157
Title: A Clinical Study Comparing Symbicort 'as Needed' With Pulmicort Twice Daily Plus Terbutaline 'as Needed' in Adult and Adolescent Patients With Asthma
Brief Title: A Clinical Study to Evaluate Symbicort Turbuhaler Used 'as Needed' in Adults and Adolescents With Asthma
Acronym: SYGMA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D589SC00003; 2013-004473-28 (EudraCT Number)
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort "as needed"+placebo Pulmicort bid (Experimental): Symbicort (budesonide/formoterol) Turbuhaler 160/4.5 μg 'as needed' + Placebo Pulmicort Turbuhaler 200 μg bid
  Interventions: Drug: budesonide/formoterol 'as needed' + budesonide placebo bid
- Pulmicort bid + terbutaline "as needed" (Active Comparator): Pulmicort 200 μg Turbuhaler bid + terbutaline 0.4 mg Turbuhaler 'as needed'
  Interventions: Drug: budesonode bid + terbutaline 'as needed'

INTERVENTIONS:
Drug: budesonide/formoterol 'as needed' + budesonide placebo bid — Symbicort (budesonide/ formoterol) 160/4.5 μg powder for inhalation 'as needed' plus Pulmicort placebo 200 μg powder for inhalation, 1 inhalation twice daily (morning and evening), 52-week treatment
  Arms: Symbicort "as needed"+placebo Pulmicort bid
Drug: budesonode bid + terbutaline 'as needed' — Pulmicort (budesonide) 200 μg powder for inhalation, 1 inhalation twice daily (morning and evening) plus terbutaline 0.4 mg powder for inhalation 'as needed', 52-week treatment
  Arms: Pulmicort bid + terbutaline "as needed"

SUMMARY:
The purpose of this study is to test if Symbicort (budesonide/formoterol) Turbuhaler is effective in treating asthma when used 'as needed' in patients with milder asthma. The efficacy of Symbicort 'as needed' will be compared with Pulmicort (budesonide) Turbuhaler twice daily plus terbutaline Turbuhaler 'as needed'

DETAILED DESCRIPTION:
A 52-week, double-blind, randomised, multi-centre, phase III, parallel-group study in patients 12 years and older with asthma, evaluating the efficacy and safety of Symbicort (budesonide/formoterol) Turbuhaler 160/4.5 μg 'as needed' compared with Pulmicort (budesonide) Turbuhaler 200 μg twice daily plus terbutaline Turbuhaler 0.4 mg 'as needed'

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures. For patients under-age, signed informed consent from both the patient and the patient's parent/legal guardian is required
2. Male or Female, ≥12 years of age
3. Documented diagnosis of asthma for at least 6 months prior to Visit 1
4. Patients who are in need of GINA step 2 treatment
5. Patients treated with a short acting inhaled bronchodilator(s) only should have pre-bronchodilator FEV1 ≥ 60 % of predicted normal (PN) and post-bronchodilator FEV1 ≥ 80 % PN
6. Patients treated with low stable dose of ICS or leukotriene antagonists in addition to short acting inhaled bronchodilator(s) should have pre-bronchodilator FEV1 ≥80 % PN
7. Patients should have reversible airway obstruction
8. To be randomized patients must have used Bricanyl Turbuhaler as needed on at least 3 separate days during the last week of the run in period

Exclusion Criteria:

1. Patient has a history of life-threatening asthma including intubation and intensive care unit admission
2. Patient has had an asthma worsening requiring change in treatment other than short acting inhaled bronchodilator(s) within 30 days prior to Visit 1 and from Visit 1 until randomization
3. Patient has required treatment with oral, rectal or parenteral GCS within 30 days and/or depot parenteral GCS within 12 weeks prior to Visit 1
4. Current or previous smoker with a smoking history of ≥ 10 pack years
5. Pregnancy, breast-feeding or planned pregnancy during the study

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4215 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, MD, Study Director — AstraZeneca Research & Development
Locations (244):
- Research Site, Sydney, Australia
- Brazil (8):
  - Research Site, Botucatu
  - Research Site, Florianópolis
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Bulgaria (13):
  - Research Site, Blagoevgrad
  - Research Site, Pernik
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Razlog
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vidin
  - Research Site, Yambol
- Chile (5):
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Viña del Mar
- Colombia (3):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Medellín
- Czechia (15):
  - Research Site, Česká Lípa
  - Research Site, Kladno
  - Research Site, Kralupy nad Vltavou
  - Research Site, Kutná Hora
  - Research Site, Liberec
  - Research Site, Neratovice
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Rudna U Prahy
  - Research Site, Tábor
  - Research Site, Teplice
  - Research Site, Žatec
- France (6):
  - Research Site, Brii-sous-forges
  - Research Site, Colmar
  - Research Site, Joué-lès-Tours
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Rezé
- Germany (16):
  - Research Site, Bad Lippspringe
  - Research Site, Berlin
  - Research Site, Cottbus
  - Research Site, Frankfurt am Main
  - Research Site, Geesthacht
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Neu-Isenburg
  - Research Site, Oldenburg
  - Research Site, Reinfeld
  - Research Site, Rüdersdorf
  - Research Site, Schleswig
  - Research Site, Warendorf
- Hungary (18):
  - Research Site, Aszód
  - Research Site, Balassagyarmat
  - Research Site, Berettyóújfalu
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Érd
  - Research Site, Gödöllő
  - Research Site, Gyula
  - Research Site, Hajdúnánás
  - Research Site, Létavértes
  - Research Site, Makó
  - Research Site, Miskolc
  - Research Site, Mórahalom
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Szeged
  - Research Site, Szombathely
  - Research Site, Vásárosnamény
- Mexico (9):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, México
  - Research Site, San Juan del Río
  - Research Site, Tlanepantla
  - Research Site, Villahermosa
  - Research Site, Zapopan
- New Zealand (12):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Christchurch Central
  - Research Site, Grafton
  - Research Site, Hamilton West
  - Research Site, Maroubra
  - Research Site, New Lambton
  - Research Site, Newtown
  - Research Site, Rotorua
  - Research Site, South Brisbane
  - Research Site, Tauranga
  - Research Site, Wellington
- Peru (5):
  - Research Site, Chancay
  - Research Site, Lima
  - Research Site, Lima Cercado
  - Research Site, Miraflores
  - Research Site, Santa Beatriz
- Philippines (4):
  - Research Site, Lipa City
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (15):
  - Research Site, Bialystok
  - Research Site, Giżycko
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Mrągowo
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Ostrów Wielkopolski
  - Research Site, Pabianice
  - Research Site, Piła
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Zabrze
- Romania (7):
  - Research Site, Bragadiru
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Deva
  - Research Site, Iași
  - Research Site, Piteşti
- Russia (23):
  - Research Site, Chelyabinsk
  - Research Site, Gatchina
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Pskov
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Ulyanovsk
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Vsevolozhsk
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Saudi Arabia (3):
  - Research Site, Dhahran
  - Research Site, Jeddah
  - Research Site, Riyadh
- Slovakia (17):
  - Research Site, Kežmarok
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Liptovský Mikuláš
  - Research Site, Lučenec
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Poprad
  - Research Site, Rimavská Sobota
  - Research Site, Ružomberok
  - Research Site, Skalica
  - Research Site, Šurany
  - Research Site, Topoľčany
  - Research Site, Trebišov
  - Research Site, Zvolen
  - Research Site, Žilina
- South Africa (10):
  - Research Site, Bellville
  - Research Site, Boksburg North
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Lenasia
  - Research Site, Mowbray
  - Research Site, Panorama
  - Research Site, Phoenix
  - Research Site, Verulam
- South Korea (9):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
- Spain (11):
  - Research Site, Alicante
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Seville
  - Research Site, Terrassa (Barcelona)
  - Research Site, Valencia
- Sweden (6):
  - Research Site, Borås
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Värnamo
  - Research Site, Västra Frölunda
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Chon Buri
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang,
  - Research Site, Nonthaburi
  - Research Site, Pathum Thani
- Ukraine (15):
  - Research Site, Cherkasy
  - Research Site, Chernihiv
  - Research Site, Chernivtsi
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kherson
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- Vietnam (6):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh
  - Research Site, Huế

REFERENCES:
- [Derived] FitzGerald JM, O'Byrne PM, Bateman ED, Barnes PJ, Zheng J, Ivanov S, Lamarca R, Larsdotter U, Emerath U, Jansen G, Puu M, Alagappan VKT, Surmont F, Reddel HK. Safety of As-Needed Budesonide-Formoterol in Mild Asthma: Data from the Two Phase III SYGMA Studies. Drug Saf. 2021 Apr;44(4):467-478. doi: 10.1007/s40264-020-01041-z. Epub 2021 Feb 6. PMID 33548020
- [Derived] Bateman ED, Reddel HK, O'Byrne PM, Barnes PJ, Zhong N, Keen C, Jorup C, Lamarca R, Siwek-Posluszna A, FitzGerald JM. As-Needed Budesonide-Formoterol versus Maintenance Budesonide in Mild Asthma. N Engl J Med. 2018 May 17;378(20):1877-1887. doi: 10.1056/NEJMoa1715275. PMID 29768147
- [Derived] O'Byrne PM, FitzGerald JM, Zhong N, Bateman E, Barnes PJ, Keen C, Almqvist G, Pemberton K, Jorup C, Ivanov S, Reddel HK. The SYGMA programme of phase 3 trials to evaluate the efficacy and safety of budesonide/formoterol given 'as needed' in mild asthma: study protocols for two randomised controlled trials. Trials. 2017 Jan 10;18(1):12. doi: 10.1186/s13063-016-1731-4. PMID 28069068
- [Derived] Reddel HK, Busse WW, Pedersen S, Tan WC, Chen YZ, Jorup C, Lythgoe D, O'Byrne PM. Should recommendations about starting inhaled corticosteroid treatment for mild asthma be based on symptom frequency: a post-hoc efficacy analysis of the START study. Lancet. 2017 Jan 14;389(10065):157-166. doi: 10.1016/S0140-6736(16)31399-X. Epub 2016 Nov 30. PMID 27912982
- See also: D589SC00003-revised-csp-edition-4_12Oct2016_Redacted_pdfa — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2649&filename=d589sc00003-revised-csp-edition-4_12Oct2016_Redacted_pdfa.pdf
- See also: D589SC00003-statistical-analysis-plan-edition-2_06SEP2017_pdfa — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2649&filename=D589SC00003-statistical-analysis-plan-edition-2_06SEP2017_pdfa.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4215 patients were enrolled. 26 patients were randomised in error and hence never recieved treatment.
Pre-assignment Details: Screening Details Eligibility was assessed at Visits 1, 2 and 3. IC was obtained at V1. At V2, patients stopped pre-study asthma medications and entered a 2 to 4 week run-in period on SABA as needed only (Bricanyl Turbuhaler 0.5 mg). Lung function was assessed by spirometry to confirm eligibility. Eligible patients were randomised at V3.
Groups:
- Placebo Bid + Symbicort 'as Needed' (Experimental): Placebo for budesonide (Placebo Turbuhaler) + Symbicort Turbuhaler (budesonide/formoterol 160/4.5 μg)
- Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator): Pulmicort Turbuhaler (budesonide 200 μg) + Terbutaline Turbuhaler 0.4mg 'as needed'
Period: Overall Study
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Started (Patients randomised and received treatment) | 2095 | 2094
Patients Who Completed Treatment | 1924 | 1903
Completed | 1985 | 1983
Not Completed | 110 | 111
Not completed — Severe non-compliance to protocol | 2 | 2
Not completed — Other | 13 | 10
Not completed — Subject decision | 58 | 50
Not completed — Prematurely closed site | 4 | 2
Not completed — Eligibility criteria not fulfilled | 4 | 8
Not completed — Lost to Follow-up | 27 | 35
Not completed — Death | 1 | 1
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator) | Total
Number analyzed (Participants) | 2089 | 2087 | 4176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (16.8) | 40.7 (17.1) | 41.0 (17.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1308 | 1289 | 2597
  Male | 781 | 798 | 1579
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    American Indian or Alaska Native | 36 | 32 | 68
    Asian | 399 | 403 | 802
    Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
    Black or African American | 34 | 33 | 67
    White | 1408 | 1406 | 2814
    Other | 211 | 211 | 422

OUTCOME MEASURES:

1. Primary Outcome: Annual Severe Asthma Exacerbation Rate - Non-inferiority Analysis
Description: Severe asthma exacerbations over the randomised treatment period, negative binomial model for non-inferiority test evaluation
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations per participant year
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
exacerbations per participant year | 0.11 [0.10 to 0.13] | 0.12 [0.10 to 0.14]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Non-Inferiority — Non-inferiority analysis based on CI instead of p-value, hence no p-value calculated for this analysis. Upper limit of the 1-sided 95% confidence limit <1.2 indicates Symbicort 'as needed' is non-inferior to Pulmicort bid; Negative binomial model; Adjusted for randomised treatment, pre-study treatment and region. Logarithm of follow-up time is used as an offset variable; Rate ratio = 0.97, 95% CI 1-sided [upper limit 1.16] — A rate ratio less than 1 indicates a lower rate of exacerbations in the Symbicort 'as needed' treatment group

2. Secondary Outcome: Number of Participants Experiencing at Least One Severe Asthma Exacerbation
Description: A severe exacerbation is defined as a deterioration of asthma requiring any of the following: use of systemic glucocorticosteroids (GCS) for at least 3 days, inpatient hospitalization, or emergency room visit due to asthma that required systemic steroids.
Time Frame: Day 1 up to 52 weeks
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
Participants | 177 | 184
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; p = 0.664, Regression, Cox; Cox regression model with randomised treatment, pre-study treatment and region as covariates; Hazard Ratio (HR) = 0.955, 95% CI 2-sided [0.777 to 1.174] — A hazard ratio less than 1 indicates that Symbicort 'as needed' prolongs the time to first severe exacerbation

3. Secondary Outcome: Average Change From Baseline in Pre-bronchodilator FEV1
Description: The average change from baseline (baseline defined by measurement at week 0, prior to first dose of IP) to the treatment period average assessed over the entire treatment period in pre-bronchodilator FEV1 was derived by computing a contrast for the mean across the post-randomisation visits (week 17, 34, 52) from the MMRM (mixed model repeated measures) analysis.
Time Frame: Study weeks 0,17, 34, 52
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
mL | 104.0 [88.5 to 119.6] | 136.6 [121.1 to 152.2]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; p = 0.003, Mixed Models Analysis; Rand treatment,pre-study treatment,region,visit,rand treatment by visit; fixed effects. Patient; random effect, baseline FEV1; covariate; Least Square Mean Difference = -32.6, 95% CI 2-sided [-53.7 to -11.4] — Mean difference greater than 0 favours Symbicort 'as needed'. Estimate corresponds to average treatment effect across all treatment visits

4. Secondary Outcome: Number of Participants With Study Specific Asthma Related Discontinuation
Description: The following two criteria lead to discontinuation from the IP due to asthma related events: A severe asthma exacerbation with duration for more than 3 weeks, and/or three severe asthma exacerbations during 6 months.
Time Frame: Day 1 up to 52 weeks
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
Participants | 0 | 4

5. Secondary Outcome: Average Change From Baseline in 'as Needed' Use
Description: 'As-needed' use change from baseline over the randomised treatment period. Baseline was defined as the last 10 days of the run-in period. 'As needed' use was calculated as the cumulative doses of 'as-needed' medication over the randomised treatment period divided by the follow-up time (number of days - 1). ie, average number of inhalations per day.
Time Frame: Week 0 up to 52 weeks
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of inhalations per day
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
Number of inhalations per day | -0.84 [-0.86 to -0.81] | -0.87 [-0.89 to -0.84]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; ANCOVA — No p-value was calculated for this efficacy variable; Model with randomised treatment, pre-study treatment and region as factors, and no. of 'as needed' inhalations at baseline as continuous covariate; Least Square Mean Difference = 0.03, 95% CI 2-sided [0.00 to 0.07] — A mean difference less than zero indicates a larger mean reduction in number of 'as needed' inhalations in the Symbicort 'as needed' group

6. Secondary Outcome: Change From Baseline in Percent of 'as Needed' Free Days
Description: 'As needed' free days (%) change from baseline during randomised treatment period. An 'as-needed' free day was defined as a day and night with no use of 'as needed' medication. Variable analysed is the percentage (%) of 'as-needed' free days during the randomised treatment period. Baseline is defined by the last 10 days of the run-in period.
Time Frame: Week 0 up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of 'as needed' free days
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
Percentage of 'as needed' free days | 41.01 [39.90 to 42.12] | 47.86 [46.75 to 48.98]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; p < 0.001, ANCOVA; adjusted for randomised treatment, pre-study treatment and region as factors and the percent 'as needed' free days during run-in as a cont covariate; Least Square Mean Difference = -6.85, 95% CI 2-sided [-8.37 to -5.34] — An estimate of difference >0 means that there was a larger increase in the % of 'as needed' free days in the Symbicort 'as-needed' arm

7. Secondary Outcome: Percentage of Controller Use Days
Description: ICS controller use days (%) during the randomised treatment period is calculated as the cumulative days when any controller medication (containing ICS) was taken including maintenance (Pulmicort bid group) and 'as needed' medication (Symbicort 'as needed' group) and additional prescribed ICS for asthma (all treatment groups), divided by the number of days in the randomised treatment period.
Time Frame: Week 0 up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
Percentage of days | 30.45 [29.20 to 31.70] | 67.92 [66.67 to 69.17]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; p < 0.001, ANOVA; model adjusted for: randomised treatment, pre-study treatment and region; Least Square Mean Difference = -37.48, 95% CI 2-sided [-39.18 to -35.77] — An estimate of difference >0 means that there was a higher % of controller use days in the Symbicort 'as-needed' group

8. Secondary Outcome: Average Change From Baseline in Asthma Control Questionnaire (5-item Version) - ACQ-5 Score
Description: ACQ questionnaire contains five questions on patients' symptoms, which are assessed on a 7-point scale from 0 (representing good control) to 6 (representing poor control). The score is the mean score of all questions for which responses are provided. The average change from baseline to treatment period average in ACQ-5 was derived by computing a contrast for the mean across all post-randomisation visits (week 17, 34, 52) from the MMRM (mixed model repeated measures) analysis.
Time Frame: Study weeks 0, 17, 34, 52
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
Score | -0.35 [-0.38 to -0.32] | -0.46 [-0.49 to -0.43]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; p < 0.001, Mixed Models Analysis; rand treatment, pre-study treatment, region, visit, rand treat by visit as fixed, patient as random, and baseline ACQ-5 as covariate; Least Square Mean Difference = 0.109, 95% CI 2-sided [0.068 to 0.150] — Mean difference less than 0 favours Symbicort 'as needed'

9. Secondary Outcome: Average Change From Baseline in Asthma Quality of Life Questionnaire Standardised Version - AQLQ(S) Score
Description: AQLQ(S) consists of 32 questions in 4 domains. Each question is assessed on a 7-point scale from 1 to 7, with higher values indicating better health-related quality of life. The overall score is calculated as the mean score of all 32 items. The average change from baseline to treatment period average in AQLQ(S) overall score was derived by computing a contrast for the mean across all post-randomisation visits (week 17, 34, 52) from the MMRM (mixed model repeated measures) analysis.
Time Frame: Study weeks 0,17, 34, 52
Population: Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: AQLQ(S) overall score
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
AQLQ(S) overall score | 0.335 [0.305 to 0.366] | 0.431 [0.400 to 0.461]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; p < 0.001, Mixed Models Analysis; rand treatment, pre-study treatment, region, visit, rand treat by visit as fixed, patient as random and baseline AQLQ as covariate; Least Square Mean Difference = -0.096, 95% CI 2-sided [-0.137 to -0.054] — Mean difference greater than 0 favours Symbicort 'as needed'

10. Primary Outcome: Annual Severe Asthma Exacerbation Rate - Superiority Analysis
Description: Severe asthma exacerbations over the randomised treatment period, negative binomial model for superiority test evaluation
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations per participant year
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
Number analyzed (Participants) | 2089 | 2087
exacerbations per participant year | 0.11 [0.10 to 0.13] | 0.12 [0.10 to 0.14]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' (Experimental) vs Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator); Test type: Superiority; p = 0.754, Negative binomial model; [statistical method as in outcome 1, analysis 1]; Rate ratio = 0.97, 95% CI 2-sided [0.78 to 1.20] — A rate ratio less than 1 indicates a lower rate of exacerbations in the Symbicort 'as needed' treatment group

ADVERSE EVENTS:
Time Frame: Adverse events were summarised from Visit 2 throughout the randomised treatment period and including the follow-up period until the last telephone follow-up, or the last contact. Serious adverse events were recorded from the time of informed consent throughout the randomised treatment period and including the folow-up period until last telephone follow-up or last contact.
Arm/Group | Placebo Bid + Symbicort 'as Needed' (Experimental) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator)
All-Cause Mortality (participants affected / at risk) | 1/2089 | 1/2087
Serious Adverse Events (participants affected / at risk) | 66/2089 | 73/2087
Other Adverse Events (participants affected / at risk) | 491/2089 | 519/2087
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Bid + Symbicort 'as Needed' (Experimental) (N=2089) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator) (N=2087)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adams-Stokes syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Degenerative aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 17 (17)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hydrocholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cystistis interstitial (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbosacral plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Bid + Symbicort 'as Needed' (Experimental) (N=2089) | Pulmicort Bid + Terbutaline 'as Needed' (Active Comparator) (N=2087)
Viral upper respiratory tract infection (Infections and infestations) | 155 (188) | 168 (206)
Asthma (Respiratory, thoracic and mediastinal disorders) | 81 (95) | 84 (96)
Headache (Nervous system disorders) | 51 (69) | 50 (68)
Bronchitis (Infections and infestations) | 64 (70) | 78 (83)
Upper respiratory tract infection (Infections and infestations) | 81 (90) | 89 (112)
Pharyngitis (Infections and infestations) | 51 (55) | 62 (74)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 51 (56) | 44 (46)
Influenza (Infections and infestations) | 33 (34) | 42 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT02224157/SAP_000.pdf
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT02224157/Prot_001.pdf